CLINICAL TRIAL: NCT04410679
Title: Treatment of Internal Inflammatory Root Resorption Using Injectable PRF Revascularization Technique: A Clinical Study With Cone Beam Computed Tomography Evaluation
Brief Title: Treatment of Internal Inflammatory Root Resorption Using Injectable PRF Revascularization Technque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mohamed Nageh, Lecturer of Endodontics, Fayoum University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FayoumU
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Root Resorption
Keywords: Pulp revascularization; injectable Platelet rich fibrin; i-PRF; root resorption; CBCT
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- injectabl PRF for treatment of internal root resorption (Experimental)
  Interventions: Biological: injectable PRF

INTERVENTIONS:
Biological: injectable PRF — blood sample and centrifuged to obtain i-PRF

SUMMARY:
Currently Endodontics looks forward for regeneration rather than repair. Regenerative endodontic therapy was limited to pulp revascularization of necrotic pulp in immature teeth , followed by mature teeth. Recently pulp revascularization technique by induction of blood clot was applied in the treatment of inflammatory root resorption. So far, no clinical study for management of teeth with inflammatory internal root resorption by using injectable PRF revascularization has been described in the literature. Thus, this is the first clinical attempt to manage inflammatory root resorption in necrotic incisor teeth using injectable PRF regenerative approach.

DETAILED DESCRIPTION:
13 teeth in a total of 10 patients with inflammatory root resorption will be treated using revascualrization technique, iPRF will be prepared and unjected in the canal after previous canal disinfection with calcium hydroxide for 2-4 weeks. cBCT will be taken preoperative and 12 month follow up period, also clinical and radiographic follow uo will be considered every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* patients 13-30 years old
* no sex predilection
* medically free
* Suffering from internal inflammatory root resorption in permanent anterior mature teeth
* associated with or without periapical radiolucency
* no or grade I tooth mobility, and a pocket depth <3 mm

Exclusion Criteria:

* old age
* Medically medically compromised patients

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-03 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
change in volumetric size of internal root resorption lesions | 12 months
  Measuring volumetric dimensions of resorption lesion pre and postoperatively using CBCT

SECONDARY OUTCOMES:
change in volumetric size of periapical lesions | 12 months
  Measuring volumetric dimensions of periapical lesion pre and postoperatively using CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Nageh, Lecturer, Principal Investigator — Faculty of dentistry, Fayoum University
Locations (1):
- Faculty of dentistry Fayoum University, Al Fayyum, Egypt